CLINICAL TRIAL: NCT06338267
Title: Validation of Innovative Biosensors for Rett Autonomic Symptom Tracking
Brief Title: Validating Innovative Biosensors for Rett Autonomic Symptom Tracking
Acronym: VIBRANT
Status: Recruiting | Type: Observational
Sponsor: Rett Syndrome Research Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SENS-102-RSRT
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Rett Syndrome
Keywords: Rett; MECP2; RTT; device; biosensor; Emerald; Vivalink; Kids O2; sensor
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main: Participants who are not in a separate interventional treatment trial
- Intervention: Participants who are also in a separate interventional treatment trial

SUMMARY:
The VIBRANT study aims to validate biosensors to objectively and directly measure symptoms in Rett syndrome and create confidence in the use of these devices in clinical trials. VIBRANT will use several FDA-cleared wearable biosensors and a non-wearable device to collect symptom data from patients with Rett syndrome for up to 9 weeks. Symptoms of interest include heart rate, breathing, sleep, blood oxygen levels, and movement. Participants will use the biosensors intermittently at home, document device use and symptom status, and will come to the clinic for 1 overnight sleep study. A cohort of up to 10 participants receiving an intervention in a separate clinical trial may also enroll and participate on a custom device schedule for up to 1 year.

The study will provide information on the feasibility and ease of use for families at home, biosensor data will be compared to data collected at the same time from the overnight sleep study to demonstrate how well they work in individuals with Rett syndrome, and Emerald will be developed to include movement as a measurable symptom.

DETAILED DESCRIPTION:
Clinical trials in Rett syndrome typically use subjective assessment scales to assess changes in symptoms. These scales require observer interpretation and can be subject to bias and placebo effect. They are often not fit for purpose, are adapted from other disorders, are not properly validated for use in Rett and therefore are not optimal tools to accurately and reliably assess symptom change.

The VIBRANT study aims to validate biosensors to objectively and directly measure symptoms in Rett syndrome and create confidence in these devices for use in clinical trials. VIBRANT will use several biosensors to collect symptom data from patients with Rett syndrome over 9 weeks. The devices under study include the FDA-cleared VV330 ECG patch for heart rate, Kids O2 pulse oximeter ring for blood oxygen levels; and the non-wearable device Emerald for sleep, breathing, and movement.

To be eligible, participants will have an MECP2 genetic variant considered causative for the disorder. Participants will come to the clinic for Screening for an eligibility assessment and will learn to use the biosensors. Participants will use the biosensors on an intermittent schedule at home for between approximately 4 to 9 weeks, depending on the device, and will come to the clinic for 1 overnight sleep study during the 9-week observation period. All devices will be used during the overnight sleep study. The data collected by the biosensors will be compared to the data collected from the overnight sleep study to demonstrate how well they work in individuals with Rett syndrome. A cohort of up to 10 participants receiving an intervention in a separate clinical trial may also enroll and participate on a custom device schedule for up to 1 year.

The goals of the study are to demonstrate FDA-cleared devices to assess heart rate, breathing, and oxygen saturation can be reliably used in Rett individuals, both adult and pediatric; determine how accurate and reliable the biosensor results are compared to the overnight sleep study, or to other FDA-cleared devices at home; to and to develop Emerald's ability to assess movement.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Rett syndrome with a causative MECP2 genetic variant
* Access to WiFi

Exclusion Criteria:

* Inability of participant to sleep alone
* prolonged absence from home
* medication use that may impact heart rate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants must have a documented genetic variant in MECP2 considered causative for Rett syndrome, must be generally healthy, able to tolerate device use.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Assess heart rate variability with Vivalink VV330 ECG patch | 4 weeks
  Use FDA-cleared Vivalink VV330 patch to directly and objectively measure heart rate parameters
Assess blood oxygen levels with Viatom Kids O2 pulse oximeter ring | 6 weeks
  Use FDA-cleared Viatom Kids O2 pulse oximeter ring to directly and objectively measure blood oxygen levels
Validate FDA-cleared Vivalink VV330 ECG patch for heart rate variability metrics in Rett syndrome compared to in-lab PSG | During PSG comparison (1 night)
  Comparison of results from ECG patch to PSG ECG results to determine accuracy and reliability
Validate ECG-derived breathing compared to in-lab PSG | During PSG comparison (1 night)
  Comparison of results from ECG-derived breathing to PSG breathing results to determine accuracy and reliability
Validate FDA-cleared Viatom Kids O2 pediatric pulse oximeter ring in Rett syndrome compared to in-lab PSG and/or Nonin wristOx pulse oximeter | During PSG comparison (1 night)
  Comparison of results from pulse oximeter ring to PSG pulse oximeter results to determine accuracy and reliability
Validate Emerald ability to reliably measure breathing and sleep compared to in-lab PSG | During PSG comparison (1 night)
  Compare Emerald to directly and objectively measure sleep and night time breathing
Validate Emerald ability to reliably measure breathing and sleep at home compared to FDA-cleared comparator | 9 weeks
  Compare Emerald to FDA-cleared SleepView home sleep test to directly and objectively measure sleep and night time breathing
Develop Emerald ability to measure daytime movement | 9 weeks
  Compare Emerald signals of movement with video

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Rush University Medical Center, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No